CLINICAL TRIAL: NCT03173443
Title: Comparison of Insertion Time Over Fiberoptic Bronchoscope Between Double Lumen Tube and Single Lumen Tube
Brief Title: Insertion Time Over Fiberoptic Bronchoscope of Double Lumen Tube and Single Lumen Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, DAE HEE KIM, Assistant Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: AJIRB-DEV-OBS-17-70
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Intubation;Difficult
Keywords: Fiberoptic intubation; double lumen tube

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single lumen tube (Experimental): fiberoptic intubation with single lumen tube with bronchial blocker.
  Interventions: Device: single lumen tube and bronchial blocker
- double lumen tube (Experimental): fiberoptic intubation with double lumen tube.
  Interventions: Device: double lumen tube

INTERVENTIONS:
Device: single lumen tube and bronchial blocker — fiberoptic intubation with single lumen tube and bronchial blocker
  Arms: single lumen tube
Device: double lumen tube — fiberoptic intubation with double umen tube
  Arms: double lumen tube

SUMMARY:
One lung ventilation (OLV) is required during thoracic procedures such as lung and esophagus surgery. three technique can be employed. (1) placement of a double-lumen bronchial tube (DLT); (2) use of a single-lumen tracheal tube (SLT) in conjunction with a bronchial blocker; (3) insertion of a conventional SLT into a main bronchus. Flexible fiberoptic intubation with SLT is well established technique for anticipated or unexpected difficult intubation. But, little is known about flexible fiberoptic intubation with DLT.

The investigators compared insertion time over fiberoptic bronchoscope between SLT with bronchial blocker and DLT in patients undergoing thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing thoracic surgery and one lung ventilation American Society of Anesthesiology Physical status 1,2

Exclusion Criteria:

* abnormality of upper airway, gastroesophageal disease, risk of aspiration, BMI > 35

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2017-08-26 (Actual); Study Completion 2017-08-26 (Actual)

PRIMARY OUTCOMES:
insertion time | at anesthesia induction
  time from insertion of bronchoscope into mouth to tube placement at trachea or bronchus

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hee Kim, M.D., Principal Investigator — Ajou unversity hospital
Locations (1):
- Ajou universiry hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No